CLINICAL TRIAL: NCT00408083
Title: A Phase IIIB, Double-Blind, Multi-Center, Randomized, Cross-Over Study to Compare 0.1 Mmol/kg of Multihance With 0.1 Mmol/kg of Magnevist for Contrast-Enhanced Magnetic Resonance Angiography(CE-MRA) of Peripheral Arteries
Brief Title: Crossover Study With MultiHance vs a Comparator for Peripheral MRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Gianpaolo Pirovano, M.D. Executive Director, Corporate Medical Development, Bracco Diagnostics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MH 127
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — gadobenic acid; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MultiHance MRI contrast agent
  Interventions: Drug: MultiHance
- 2 (Active Comparator): Magnevist contrast agent for MRA
  Interventions: Drug: Magnevist

INTERVENTIONS:
Drug: MultiHance — 0.5 mmol/kg as a single dose administration
  Arms: 1
Drug: Magnevist — 0.5 mmol/kg as a single dose administration
  Arms: 2

SUMMARY:
This is a double blind crossover study designed to compare two different gadolinium products given at the same dose to patients undergoing MRA assessment of lower legs for the evaluation of peripheral steno-occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* At least 18 yrs of age
* Moderate to severe peripheral arterial disease
* Willing to undergo two MRA procedures within 14 days

Exclusion Criteria:

* Pregnant or lactating
* Known allergies to one or more ingredients in the products
* Therapeutic intervention in the arterial territory of interest between the two MRA exams
* Changes in symptoms between the two exams
* Vascular stent in area of interest
* Severe claustrophobia
* Congestive heart failure class IV
* Scheduled to undergo surgery for PAOD between the two exams
* Scheduled to undergo DSA between the two exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assessment of global paired diagnostic preference of the two MRA exams | Post dose

SECONDARY OUTCOMES:
To compare the two different products for signal intensity enhancement; average quality of visualization; technical failure rate; to assess inter-reader agreement in terms of average quality of visualization | post dose

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Imaging, Milan, Italy